CLINICAL TRIAL: NCT05579613
Title: Faculty of Physical Therapy, Cairo University, Egypt
Brief Title: Effect of Interactive Virtual Reality Device on Cervical Proprioception and Range of Motion in Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibtsam Abdelkarim, Faculty of physical therapy, Cairo university, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003549
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes assessors will be blinded to the intervention the group wil receivee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive virtual reality device group (Experimental): Group A will receive the same as group "B" and will receiveVR training by Xbox Kinect 360 (15 min per session 3 times per week) for 4 weeks. C
  Interventions: Device: Interactive virtual reality device
- chin tuck exercise for posture correction (traditional treatment ) group (Experimental): Group B will receive traditional treatment (chin tuck exercise for posture correction); 3 min each day for 4 weeks, three sets of 10 repetitions (each repetition was held for 5 sec) will be performed.
  Interventions: Device: Interactive virtual reality device

INTERVENTIONS:
Device: Interactive virtual reality device — The Kinect sensor is an infrared camera that can recognize the positions and motions of the player without the need for special controller. The console controls the various games .For the VR training, the Xbox Kinect, console, and monitor will set up in a dedicated space. The patient will placed 1.5-2 m away from the Kinect sensor.

SUMMARY:
Forward head posture (FHP) is one of the most common postural deformities, which affects 66% of the patient population and this study will be designed to investigate the effect of interactive virtual reality device on cervical proprioception and range of motion in symptomatic forward head posture.

DETAILED DESCRIPTION:
Thirty subjects of both sex with ages ranging from 20-24 years and BMI ranging from 18-25 kg/m² with symptomatic forward head posture will be participated in this study. They will be assigned randomly to two groups. Group A will receive traditional treatment (chin tuck exercise for posture correction); 3 min each day for 4 weeks, three sets of 10 repetitions (each repetition was held for 5 sec) were performed. Group B will receive the same as group "A" and received VR training by Xbox Kinect 360 (15 min per session 3 times per week) for 4 weeks. Cervical joint position error (JPE) (CROM device) and cervical range of motion will be measured pre and post treatment.

ELIGIBILITY:
Inclusion Criteria :

1. Subject's age range from 18-24 years old distance of ≥ 2 cm between the acromion and the earlobe when they were positioned perpendicular to the ground.( Kim et al 2018).
2. Prolonged neck pain for more than three months; and the Neck Disability

Exclusion Criteria:1- Existing vestibular pathology.

2- Cervical fracture/dislocation. 3- Sys- temic diseases. 4- Neurological/cardiovascular/respiratory disorders affecting physical performance.

5- History of traumatic head injury. 6- Pregnancy.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-10-03 (Estimated)

PRIMARY OUTCOMES:
Cervical propriception | 4 weeks
  Assessment of cervical proprioception using cervical range of motion
Cervical range of motion | 4 weeks
  Assessment of cervical range of motion by CROM

CONTACTS AND LOCATIONS:
Locations (1):
- Ibtsam Abdelkarim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided